CLINICAL TRIAL: NCT01768676
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Multicenter Clinical Trial of the Effect of Avanafil (STENDRA™) on Spermatogenesis in Healthy Adult Males and Adult Males With Mild Erectile Dysfunction
Brief Title: Study Evaluating the Effects of Avanafil on Semen Parameters
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VIVUS LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TA-401
Record Dates: First submitted 2013-01-11; First posted 2013-01-15 (Estimated); Results first posted 2015-12-14 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-11

CONDITIONS: Erectile Dysfunction
Keywords: healthy male
MeSH Terms: conditions — Erectile Dysfunction | interventions — avanafil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- avanafil (Experimental): 100 mg
  Interventions: Drug: avanafil
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: avanafil — 100 mg
  Other Names: TA-1790; Stendra
  Arms: avanafil
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether avanafil will affect different aspects of sperm production.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent
* Able to produce semen samples without requiring therapy (PDE5 inhibitors, over-the-counter (OTC) medication, and/or herbal supplements) for erectile dysfunction
* Be medically healthy (no clinically significant screening results for medical history, electrocardiogram (ECG), laboratory studies, physical examination, etc.) in the opinion of the investigator
* Be willing and able to comply with all study requirements

Exclusion Criteria:

* An International Index of Erectile Function (IIEF) erectile function domain score of less than 17;
* History of infertility, vasectomy, testicular mass, testicular trauma, testicular abnormality (including size), radiation to the testis, previous pelvic surgery, cryotherapy of the prostate, known sperm defect, or retrograde ejaculation, or cryptorchidism;
* Resting heart rate <45 or >90 beats per minute at screening (3 rechecks permitted);
* Screening systolic blood pressure <90 or >140 mmHg and/or diastolic blood pressure <50 or >90 mmHg (3 rechecks permitted);
* High serum FSH (>18.0 mIU/mL), high serum LH (>18 mIU/mL), or low serum testosterone (< 270 ng/dL, early morning collection) on screening;
* AST or ALT >2.0 x ULN or other evidence of significant hepatic impairment;
* Prostate specific antigen (PSA) level ≥4 ng/mL at screening;
* Individuals who perform rotating shift work during the course of the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 181 (Actual)
Dates: Start 2012-12; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Research Facility, Huntsville, Alabama
  - Research Facility, Los Angeles, California
  - Research Facility, San Diego, California
  - Research Facility, Parker, Colorado
  - Research Facility, Aventura, Florida
  - Research Facility, Carmel, Indiana
  - Research Facility, New Orleans, Louisiana
  - Research Facility, Shreveport, Louisiana
  - Research Facility, Kansas City, Missouri
  - Research Facility, Albany, New York
  - Research Facility, New York, New York
  - Research Facility, Cincinnati, Ohio
  - Research Facility, Bala-Cynwyd, Pennsylvania
  - Research Facility, Knoxville, Tennessee
  - Research Facility, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Avanafil: 100 mg once daily in the evening
- Placebo: placebo taken once daily in the evening
Period: Overall Study
Arm/Group | Avanafil | Placebo
Started | 90 | 91
Completed | 66 | 60
Not Completed | 24 | 31
Not completed — Adverse Event | 3 | 3
Not completed — Lost to Follow-up | 13 | 16
Not completed — Protocol Violation | 1 | 1
Not completed — Physician Decision | 4 | 1
Not completed — Withdrawal by Subject | 3 | 10

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- Total: Total of all reporting groups
Arm/Group | Avanafil | Placebo | Total
Number analyzed (Participants) | 90 | 91 | 181
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.8 (7.23) | 32.9 (7.11) | 33.8 (7.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 90 | 91 | 181
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 29 | 53
  Not Hispanic or Latino | 66 | 62 | 128
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 28 | 16 | 44
  White | 59 | 71 | 130
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 90 | 91 | 181
Baseline sperm concentration [Mean (Standard Deviation); unit: million sperm/mL] | 76.1 (43.05) | 76.3 (40.65) | 76.2 (41.75)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With a Greater Than or Equal to 50% Decrease in Sperm Concentration From Baseline to Week 26
Description: Subjects provided 2 semen samples at each visit 2 to 12 days apart. The average value is used as the visit result.
Time Frame: Baseline to Week 26
Population: Completer population is defined as those who completed the study through week 26 and had semen analysis at both baseline and week 26. This may differ from the definition of completers for the study flow.
Measure: Number; unit: percentage of participants
Arm/Group | Avanafil | Placebo
Number analyzed (Participants) | 68 | 69
percentage of participants | 1.5 | 14.5
Statistical Analysis 1: Comparison: Avanafil vs Placebo; Test type: Non-Inferiority or Equivalence — The difference in percentage of subjects with a >/= 50% reduction from baseline to Week 26 in sperm concentration between treatment arms was analyzed using Cochran-Mantel-Haenszel method to account for the randomization stratification by baseline sperm concentration. If upper limit of 95% CI < 20% then avanafil is considered non-inferior to placebo; Risk Difference (RD) = -12.93, 95% CI 2-sided [-21.56 to -4.29], Standard Error of Mean 4.41 — Confidence interval was only calculated for primary endpoint of the difference between avanafil and placebo, not for each individual arm

2. Secondary Outcome: Percentage of Subjects With Greater Than or Equal to 50% Reduction in Sperm Count From Baseline to Week 26
Time Frame: baseline to week 26
Population: completers population
Measure: Number; unit: percentage of participants
Arm/Group | Avanafil | Placebo
Number analyzed (Participants) | 68 | 69
percentage of participants | 10.3 | 21.7
Statistical Analysis 1: Comparison: Avanafil vs Placebo; Test type: Non-Inferiority or Equivalence — If upper limit of 95% CI < 20% then avanafil is considered non-inferior to placebo; Risk Difference (RD) = -11.4, 95% CI 2-sided [-23.5 to 0.7], Standard Error of Mean 6.2 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage of Subjects With Greater Than or Equal to 50% Reduction in Sperm Motility From Baseline to Week 26
Description: Sperm motility was based upon the WHO grading scale: grade A, B, or C.
Time Frame: baseline to week 26
Population: completers population
Measure: Number; unit: percentage of participants
Arm/Group | Avanafil | Placebo
Number analyzed (Participants) | 68 | 69
percentage of participants | 0 | 1.4
Statistical Analysis 1: Comparison: Avanafil vs Placebo; Test type: Non-Inferiority or Equivalence — If upper limit of 95% CI < 20% then avanafil is considered non-inferior to placebo; Risk Difference (RD) = -1.4, 95% CI 2-sided [-4.2 to 1.3], Standard Error of Mean 1.4 — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Percentage of Subjects With Greater Than or Equal to 50% Reduction in Semen Volume From Baseline to Week 26
Time Frame: baseline to week 26
Population: completers population
Measure: Number; unit: percentage of participants
Arm/Group | Avanafil | Placebo
Number analyzed (Participants) | 68 | 69
percentage of participants | 0 | 2.9
Statistical Analysis 1: Comparison: Avanafil vs Placebo; Test type: Non-Inferiority or Equivalence — If upper limit of 95% CI < 20% then avanafil is considered non-inferior to placebo; Risk Difference (RD) = -2.9, 95% CI 2-sided [-6.8 to 1.1], Standard Error of Mean 2 — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Percentage of Subjects With Greater Than or Equal to 50% Reduction in Normal Sperm Morphology From Baseline to Week 26
Time Frame: baseline to week 26
Population: completers population
Measure: Number; unit: percentage of participants
Arm/Group | Avanafil | Placebo
Number analyzed (Participants) | 68 | 69
percentage of participants | 0 | 0
Statistical Analysis 1: Comparison: Avanafil vs Placebo; Test type: Non-Inferiority or Equivalence — If upper limit of 95% CI < 20% then avanafil is considered non-inferior to placebo; Risk Difference (RD) = 0, 95% CI 2-sided [0 to 0], Standard Error of Mean 0 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Arm/Group | Avanafil | Placebo
Serious Adverse Events (participants affected / at risk) | 0/90 | 1/91
Other Adverse Events (participants affected / at risk) | 14/90 | 20/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avanafil (N=90) | Placebo (N=91)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avanafil (N=90) | Placebo (N=91)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2)
Tooth abscess (Infections and infestations) | 0 (0) | 2 (3)
abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 3 (7)
Bronchititis (Infections and infestations) | 1 (1) | 0 (0)
rhinitis (Infections and infestations) | 1 (1) | 0 (0)
upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
influenza (Infections and infestations) | 0 (0) | 1 (1)
periodontitis (Infections and infestations) | 0 (0) | 1 (1)
pilonidal cyst (Infections and infestations) | 0 (0) | 1 (1)
urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
hyperaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
flushing (Vascular disorders) | 1 (1) | 0 (0)
hot flush (Vascular disorders) | 1 (1) | 0 (0)
hypertension (Vascular disorders) | 1 (1) | 0 (0)
pain (General disorders) | 1 (1) | 0 (0)
decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
premature ejaculation (Psychiatric disorders) | 1 (1) | 0 (0)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
palpitations (Cardiac disorders) | 0 (0) | 1 (1)
nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
semenuria (Renal and urinary disorders) | 0 (0) | 1 (1)
urethral meatus stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
urinary straining (Renal and urinary disorders) | 0 (0) | 1 (1)
urine flow decreased (Renal and urinary disorders) | 0 (0) | 1 (1)
penis disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1)
testicular disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1)
acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After Sponsor's written notification that publication of results is no longer planned or 12 months after termination of the study at all sites, Institution & PI may publish, upon written approval from Sponsor, results of the Study. Sponsor will be given the opportunity to review any proposed publication at least 60 days prior to submission for publication or disclosure. Upon Sponsor's written request, Institution and PI shall not publish or disclose information related to the Study.